CLINICAL TRIAL: NCT06797934
Title: Establishment of a Registry of Patients With Parathyroid Disease
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PARAT
Record Dates: First submitted 2024-12-03; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-11

CONDITIONS: Hyperparathyroidism; Hypoparathyroidism
MeSH Terms: conditions — Hyperparathyroidism; Hypoparathyroidism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Establishment of a registry with which to census all patients under the care of the O.U. Endocrinology for parathyroid pathology in order to longitudinally evaluate biochemical, clinical, radiological, medico-nuclear and histological data in future studies.

DETAILED DESCRIPTION:
Inclusion in the registry will be offered consecutively to any patient with parathyroid pathology (hyperparathyroidism or hypoparathyroidism) diagnosed and evaluated at the Endocrinology Operating Unit through at least two endocrinology visits. The registry will include patients seen from 1/1/2000 for a duration of 30 years. Follow-up duration for each patient is expected to be 10 years, with enrollment until 12/31/2029, and registry update deadline on 12/31/2039.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of hyperparathyroidism or hypoparathyroidism based on biochemical parameters (calcemia, parathormone, phosphormia, creatinine, albumin, vitamin D25OH)
* Obtaining informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion in the registry will be offered consecutively to any patient with parathyroid pathology (hyperparathyroidism or hypoparathyroidism) diagnosed and evaluated at the Endocrinology Operating Unit through at least two endocrinology visits. The registry will include patients seen from 1/1/2000 for a duration of 30 years. Follow-up duration for each patient is expected to be 10 years, with enrollment until 12/31/2029, and registry update deadline on 12/31/2039.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2039-12-30 (Estimated); Study Completion 2039-12-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal Biochemical Monitoring in Patients with Parathyroid Pathology | through study completion, an average of 15 years
  This outcome measure will specifically assess and report biochemical parameters in patients with parathyroid pathology under the care of the O.U. Endocrinology. Key biochemical markers to be measured include:
  Serum calcium levels (mmol/L) Serum phosphorus levels (mmol/L) Parathyroid hormone (PTH) levels (pg/mL) Vitamin D levels (ng/mL) Each parameter will be measured at baseline and at predefined intervals throughout the study. The collected data will be summarized as means ± standard deviations for continuous variables or as proportions for categorical data, where appropriate.
Clinical Outcomes in Parathyroid Pathology: Symptom Severity, Biochemical Parameters, and Comorbidities | through study completion, an average of 15 years
  This outcome measure includes the assessment of multiple clinical parameters related to parathyroid pathology. These include:
  Symptom Severity: Assessed using a standardized symptom severity scale, reported as a score.
  Biochemical Parameters: Measurement of serum calcium levels (mg/dL) and parathyroid hormone (PTH) levels (pg/mL), summarized as means ± standard deviation.
  Comorbidities: Documented as binary variables (present/absent) and reported as prevalence percentages.
Radiological Assessments in Parathyroid Pathology: Imaging Findings and Anatomical Evaluation | through study completion, an average of 15 years
  This outcome measure involves the collection and evaluation of radiological data to assess the anatomical and functional status of the parathyroid glands and related structures. Specific assessments include:
  Ultrasound Findings: Measurement of gland size (in centimeters) and structural abnormalities.
  CT and MRI Results: Detection of anatomical changes or lesions, reported as present/absent and described qualitatively.
  Bone Scans: Evaluation of bone metabolism abnormalities, summarized as binary outcomes (normal/abnormal).
  Each imaging modality will be analyzed and reported independently, with results summarized based on specific Units of Measure, such as size (cm) or qualitative descriptors.
Medico-Nuclear Outcomes: Parathyroid Imaging and Functional Assessment | through study completion, an average of 15 years
  This outcome measure focuses on data obtained from nuclear medicine imaging to evaluate parathyroid gland function. Specific assessments include:
  Sestamibi Scan Results: Reported as qualitative findings (e.g., positive/negative for abnormal uptake) and quantified when applicable (e.g., uptake percentage).
  Additional Imaging Modalities: Data from parathyroid-specific imaging (e.g., PET/CT or ultrasound) will include quantitative parameters such as gland size (cm³) and uptake intensity scores.
  Each imaging modality will be analyzed and reported separately using appropriate Units of Measure. Aggregation methods will be clarified if data from multiple imaging types are combined to inform a single outcome metric.
Histopathological Characteristics of Parathyroid Pathology | through study completion, an average of 15 years
  This outcome measure focuses on the collection and analysis of histological data from tissue samples. Specifically:
  Biopsy Results: Histopathological features will be described qualitatively (e.g., presence of adenoma, hyperplasia) and quantitatively (e.g., cell counts, mitotic index per high-power field).
  Post-Surgical Tissue Analysis: Includes structural characteristics such as tissue size (measured in millimeters), cellular composition, and presence of fibrosis or calcifications.
  Each type of histopathological finding will be documented and analyzed independently, with appropriate Units of Measure used for quantitative assessments. Aggregated data will be summarized to provide insights into the cellular and structural characteristics of parathyroid pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Uberto Pagotto, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No